CLINICAL TRIAL: NCT01099475
Title: Randomized Controlled Trial on the Effect of Intermittent Pedicle Clamping Using 15 or 30 Minutes Ischemic Intervals During Liver Surgery
Brief Title: Effect of Intermittent Pedicle Clamping on Hepatocellular Injury During Liver Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 06-2-067
Record Dates: First submitted 2010-04-01; First posted 2010-04-07 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Hepatocellular Injury; Blood Loss
Keywords: liver surgery; pringle manoeuvre; hepatocellular damage; surgical complications; patients requiring liver surgery
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pringle manoeuvre 15 minutes (Experimental): When intermittent pedicle occlusion during parenchymal transection is necessary, 2 cycles of 15 minutes of hepatic inflow occlusion will be applied each followed by 5 minutes of reperfusion. During inflow occlusion, the complete portal triad was clamped using a rubber sling.
  Interventions: Procedure: Pringle manoeuvre 15 minutes
- Pringle manoeuvre 30 minutes (Experimental): When intermittent pedicle occlusion during parenchymal transection is necessary, 1 cycle of 30 minutes of hepatic inflow occlusion will be applied followed by 5 minutes of reperfusion. During inflow occlusion, the complete portal triad was clamped using a rubber sling.
  Interventions: Procedure: Pringle manoeuvre 30 minutes

INTERVENTIONS:
Procedure: Pringle manoeuvre 15 minutes — During parenchymal transection, the hepatoduodenal ligament will be clamped by a rubber band for 2-times 15 minutes with 5 minutes reperfusion
  Arms: Pringle manoeuvre 15 minutes
Procedure: Pringle manoeuvre 30 minutes — During parenchymal transection, the hepatoduodenal ligament will be clamped by a rubber band for 30 minutes with 5 minutes reperfusion
  Arms: Pringle manoeuvre 30 minutes

SUMMARY:
In order to prevent excessive blood loss during liver surgery, an intermittent Pringle manoeuvre (IPM) can be applied. This implies a temporary clamping of the portal vein and hepatic artery in the hepatoduodenal ligament in order to occlude hepatic inflow. The optimal duration of the IPM is unknown. This randomized controlled trial aimed to analyse differences in hepatocellular damage after 15 minutes or 30 minutes IPM during liver surgery for primary or secondary liver tumours.

DETAILED DESCRIPTION:
Surgical procedure Patients were anaesthetized using isoflurane and propofol. They routinely had an epidural catheter, urinary catheter, two peripheral venous catheters and indwelling catheters in a jugular vein and radial artery. Body temperature was maintained using a Bair Hugger system (Arizant Healthcare Inc. Eden Prairie, Minnesota).

The surgical procedure was performed using a subcostal bilateral incision and Olivier retractors to improve exposure. After dissection of the teres hepatis ligament, the liver was mobilized. Thereafter, an intra-operative ultrasound was performed to define the position of the tumour in relation to vascular and biliary structures. As IPM was not routinely applied, a patient was randomized for 15 minted IPM (15IPM) or 30 minutes IPM (30IPM) only after the surgeon had decided a complete Pringle manoeuvre would be required. During 15IPM or 30IPM, the complete portal triad was clamped using a rubber sling. The time of inflow occlusion was adapted to the need according to the randomization protocol. Occasionally, the left or right pedicle was ligated after protocolled IPM. Five minutes reperfusion intervals were applied during which transection was stopped and cut surfaces were gently compressed to ensure hemostasis. A Cavitron Ultrasonic Surgical Aspirator (CUSA system 200 macrodissector, Cavitron Surgical Systems, Stamford, Connecticut) and Argon beam coagulation (Force GSU System, Valleylab, Boulder, Colorado) were used for liver transection. A stapler device or clamps were used for transection of the hepatic veins. Central venous pressure was maintained below 5 centimetre of water (cm H2O) during transection to reduce venous back-bleeding. After surgery, the weight of the resection specimen was recorded. Perioperative care was protocolled, as described earlier.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years of age and < 100 years of age
* primary or secondary liver tumours requiring liver surgery

Exclusion Criteria:

* pre-existent liver disease (e.g. inflammatory liver disease, cirrhosis, inborn errors of metabolism)
* cholangiocarcinoma requiring biliary tract reconstruction during surgery
* steroid hormone medication
* tumours deemed irresectable during liver surgery
* laparoscopic liver surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis HC Dejong, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, PO Box 5800, Netherlands

REFERENCES:
- [Result] van den Broek MA, Bloemen JG, Dello SA, van de Poll MC, Olde Damink SW, Dejong CH. Randomized controlled trial analyzing the effect of 15 or 30 min intermittent Pringle maneuver on hepatocellular damage during liver surgery. J Hepatol. 2011 Aug;55(2):337-45. doi: 10.1016/j.jhep.2010.11.024. Epub 2010 Dec 13. PMID 21147188
- [Result] Dello SA, Reisinger KW, van Dam RM, Bemelmans MH, van Kuppevelt TH, van den Broek MA, Olde Damink SW, Poeze M, Buurman WA, Dejong CH. Total intermittent Pringle maneuver during liver resection can induce intestinal epithelial cell damage and endotoxemia. PLoS One. 2012;7(1):e30539. doi: 10.1371/journal.pone.0030539. Epub 2012 Jan 24. PMID 22291982

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion of participants: Oct 2007 - Jul 2009 Location: Department of Surgery, Maastricht University Medical Centre
Groups:
- Pringle Manoeuvre Using 15 Minutes Inflow Occlusion: When intermittent pedicle occlusion during parenchymal transection is necessary, 2 cycles of 15 minutes of hepatic inflow occlusion will be applied each followed by 5 minutes of reperfusion.
  Pringle manoeuvre using 15 minutes ischemic interval: During parenchymal transection, the hepatoduodenal ligament will be clamped by a rubber band for 2-times 15 minutes with 5 minutes reperfusion
- Pringle Manoeuvre Using 30 Minutes Inflow Occlusion: When intermittent pedicle occlusion during parenchymal transection is necessary, 1 cycle of 30 minutes of hepatic inflow occlusion will be applied followed by 5 minutes of reperfusion
  Pringle Manoeuvre using 30 minutes ischemic interval: During parenchymal transection, the hepatoduodenal ligament will be clamped by a rubber band for 30 minutes with 5 minutes reperfusion
Period: Overall Study
Arm/Group | Pringle Manoeuvre Using 15 Minutes Inflow Occlusion | Pringle Manoeuvre Using 30 Minutes Inflow Occlusion
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pringle Manoeuvre Using 15 Minutes Inflow Occlusion | Pringle Manoeuvre Using 30 Minutes Inflow Occlusion | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 64 [48 to 80] | 62 [30 to 77] | 62 [30 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  Netherlands | 10 | 10 | 20
American Society of Anesthesiologists (ASA) classification [Number; unit: participants] — The ASA (American Society of Anesthesiologists) physical status classification system is a system for assessing the fitness of cases before surgery and consists of a six-category physical status classification system. These are:
  ASA 1. Healthy person. ASA 2. Mild systemic disease. ASA 3. Severe systemic disease. ASA 4. Severe systemic disease that is a constant threat to life. ASA 5. A moribund person who is not expected to survive without the operation. ASA 6. A declared brain-dead person whose organs are being removed for donor purposes
  participants
    ASA 1 | 0 | 2 | 2
    ASA 2 | 8 | 5 | 13
    ASA 3 | 2 | 3 | 5
Indication for resection [Number; unit: participants]
  benign disease | 0 | 1 | 1
  malignant disease | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Hepatocellular Damage Reflected by Liver Fatty-acid Binding Protein (L-FABP) Levels
Description: At specific time points before, during and after liver surgery, plasma samples will be obtained to analyse the amount of hepatocellular damage reflected by L-FABP) level. These timepoints include: baseline (before operation), just before intermittent pedicle clamping, just before end of 15 or 30 minutes pedicle clamping, end of 5 minutes reperfusion, end of liver surgery, 8 hours after start liver surgery, postoperative day 1, 2 and 3. This continuous variable with repeated measurements was summarized as area under the curve (AUC) from baseline to postoperative day 3 (as described in Matthews JN, Altman DG, Campbell MJ, Royston P. Analysis of serial measurements in medical research. Bmj 1990;300:230-5).
Time Frame: L-FABP area under curve from start of surgery up until postoperative day 3
Measure: Mean (Standard Error); unit: ng*h/mL
Arm/Group | Pringle Manoeuvre Using 15 Minutes Inflow Occlusion | Pringle Manoeuvre Using 30 Minutes Inflow Occlusion
Number analyzed (Participants) | 10 | 10
ng*h/mL | 9097 (1781) | 11,688 (2247)

2. Secondary Outcome: Post-resectional Complications
Description: morbidity and mortality occuring after liver surgery graded according to Clavien-Dindo's grading system. In short, any deviation from the postoperative course without the need for pharmacological, radiological or surgical intervention was classified as Clavien-Dindo grade 1; complications requiring pharmacological treatment were graded as grade 2; complications requiring surgical or radiological intervention not under general anesthesia as grade 3a and under general anesthesia as grade 3b; grade 4 complications were life-threatening complications requiring intensive care unit care because of single organ dysfunction (grade 4a) or multiple organ dysfunction (grade 4b); mortality was classed as grade 5.
Time Frame: within 90-days after initial liver surgery
Measure: Number; unit: participants
Arm/Group | Pringle Manoeuvre Using 15 Minutes Inflow Occlusion | Pringle Manoeuvre Using 30 Minutes Inflow Occlusion
Number analyzed (Participants) | 10 | 10
participants
  intra-abdominal abscess | 3 | 2
  intra-abdominal hemorrhage | 0 | 1
  bile leakage | 4 | 1
  ascites | 1 | 0
  sepsis | 1 | 2
  post-resectional liver failure | 2 | 1
  30-day mortality | 1 | 1

3. Secondary Outcome: Amount of Blood Loss
Description: amount of blood in the suction container (and, if applicable, in the weighted gauzes)
Time Frame: at the end of liver surgery, an average of 225 minutes
Measure: Median (Full Range); unit: mL
Arm/Group | Pringle Manoeuvre Using 15 Minutes Inflow Occlusion | Pringle Manoeuvre Using 30 Minutes Inflow Occlusion
Number analyzed (Participants) | 10 | 10
mL | 575 [100 to 2300] | 450 [250 to 1000]

4. Secondary Outcome: Hepatocellular Damage Reflected by Alanine Aminotransferase (ALAT) Levels
Description: At specific time points before, during and after liver surgery, plasma samples will be obtained to analyse the amount of hepatocellular damage reflected by ALAT level. These timepoints include: baseline (before operation), just before intermittent pedicle clamping, just before end of 15 or 30 minutes pedicle clamping, end of 5 minutes reperfusion, end of liver surgery, 8 hours after start liver surgery, postoperative day 1, 2 and 3.
Time Frame: ALAT area under curve from start of surgery up until postoperative day 3
Measure: Mean (Standard Error); unit: IU*h/L
Arm/Group | Pringle Manoeuvre Using 15 Minutes Inflow Occlusion | Pringle Manoeuvre Using 30 Minutes Inflow Occlusion
Number analyzed (Participants) | 10 | 10
IU*h/L | 3196 (797) | 3609 (812)

ADVERSE EVENTS:
Time Frame: Reported adverse events (AE) were scored from day 0 up to day 30 after liver surgery
Arm/Group | Pringle Manoeuvre Using 15 Minutes Inflow Occlusion | Pringle Manoeuvre Using 30 Minutes Inflow Occlusion
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No